CLINICAL TRIAL: NCT01433120
Title: Targeting the Gut Microbiome to Investigate the Pathways of Progression From Obesity to Metabolic Diseases in an At-risk Population.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Lundbeck Foundation (Other); Arla Foods (Industry)
Responsible Party: Principal Investigator, Arne Astrup, MD, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-244 LuCamp
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obesity; Insulin resistance; Microbiota; Probiotic; Prebiotic
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probiotic L. casei F19 (Experimental)
  Interventions: Dietary Supplement: Lactobacillus paracasei ssp paracasei F19
- Flax seed fibres (Experimental)
  Interventions: Dietary Supplement: Flax seed fibres
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin (Placebo)

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei ssp paracasei F19 — 10^10 CFU of Lactobacillus paracasei F19 (dissolved in a glass of water once per day)
  Arms: Probiotic L. casei F19
Dietary Supplement: Flax seed fibres — 10 grams of flax seed fibres per day (baked into two breakfast buns)
  Arms: Flax seed fibres
Dietary Supplement: Maltodextrin (Placebo) — Maltodextrin is dissolved in a glas of water once per day
  Arms: Placebo

SUMMARY:
Studies of the human gut microbiome have suggested that treatment or prevention aimed at the obese microbiome could influence the development of obesity-associated metabolic disturbances.

The objective of this project is to explore if a dietary intervention in 60 obese women with the probiotic Lactobacillus paracasei ssp paracasei F19 or flax seed fibres targeting the gut microbiome, can reduce insulin resistance, low-grade inflammation or dyslipidaemia, and to explore the interaction between the human genome and the gut microbiome.

The study is based on the following hypotheses:

* Treatment with the probiotic Lactobacillus paracasei ssp paracasei F19 and flax seed fibres will lower the metabolic risk profile in the intervention groups compared with placebo.
* The effect on the metabolic risk markers can be correlated with changes in the gut microbiota (measured in faeces).

After completion of the dietary intervention, the participants are offered a 10-week weight reduction program. Those who participate in the weight-loss program are invited to an optional follow-up visit in connection with the last visit at the clinical dietician, for the purpose of exploring the effect of weight loss on the gut microbiota and obesity-associated metabolic disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal
* BMI between 30-45 kg/m2
* Waist circumference > 80 cm
* High leukocyte count

Exclusion Criteria:

* Medically-treated Type 2 diabetes or dyslipidaemia
* Use of antibiotics during the last 3 months
* Use of pro- or prebiotic supplements during the last 6 weeks
* Illnesses related to the gastro-intestinal tract
* History of psychiatric diseases (incl. depression)
* Liver disease
* Alcohol abuse

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | Week 0,6
  3H OGTT (75g glucose)
Changes in the gut microbiota | Week 0,6

SECONDARY OUTCOMES:
Inflammatory markers | Week 0,4,6
Lipid metabolism | Week 0,6
Total fat mass and abdominal fat | Week 0,6

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, MD, Professor, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (1):
- Department of Human Nutrition, Faculty of Life Sciences, University of Copenhagen, Frederiksberg C, Denmark

REFERENCES:
- See also: Related Info — http://www.lucamp.org
- See also: Related Info — http://www.ihe.life.ku.dk